CLINICAL TRIAL: NCT06068868
Title: A Phase 1 First-in-Human Study Evaluating Safety, Pharmacokinetics and Efficacy of ABBV-787 in Adult Subjects With Acute Myeloid Leukemia (AML)
Brief Title: Study to Evaluate Adverse Events and Movement of Intravenously (IV) Infused ABBV-787 in Adult Participants With Relapsed/Refractory (R/R) Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M23-477; 2023-505233-27-00 (Other: EU CT)
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML; ABBV-787
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ABBV-787 (Experimental): Participants will receive increasing doses of ABBV-787 until the maximum tolerated dose (MTD) during the 3 year treatment period.
  Interventions: Drug: ABBV-787

INTERVENTIONS:
Drug: ABBV-787 — Intravenous (IV) Infusion

SUMMARY:
Acute myeloid leukemia (AML) is the second most common type of leukemia diagnosed in adults and children, but most cases occur in adults. This study is to evaluate how safe ABBV-787 is and how it moves within the body in adult participants with relapsed/refractory (R/R) acute myeloid leukemia (AML). Adverse events and maximum tolerated dose (MTD) of ABBV-787 will be assessed.

ABBV-787 is an investigational drug being developed for the treatment of AML. Participants will receive ABBV-787 in escalating doses until the maximum tolerated dose (MTD) is determined. Approximately 60 adult participants with a diagnosis of AML will be enrolled worldwide.

Participants will receive intravenous (IV) infusions of ABBV-787 during the approximately 3 year duration a participant is followed.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Laboratory Criteria matching those outlined in the protocol.
* QT interval corrected for heart rate (QTc) <= 470 msec using Fridericia's correction, and no other clinically significant cardiac abnormalities.
* Documented diagnosis of non-promyelocytic acute myeloid leukemia (AML), per 2022 European Leukemia Net (ELN) criteria.
* Participants with relapsed/refractory (R/R) acute myeloid leukemia (AML) who have been treated with up to 3 prior lines of therapy and are refractory to or intolerant of all established AML therapies that are known to clearly provide clinical benefit at the judgement of the investigator.
* Must have a white blood cell (WBC) count < 25 × 10^9 /L prior to initiation of study drug (Note: Hydroxyurea or leukapheresis is permitted to meet this criterion and for use through Cycle 3 to control for hyperleukocytosis.).

Exclusion Criteria:

* Have received a CD33-targeting therapy within 3 months prior to the first dose of ABBV-787.
* Stem cell transplant within 3 months prior to first dose of study drug.
* Have received anticancer therapy including chemotherapy, radiation therapy, immunotherapy, biologic, or any investigational therapy within 14 days or 5 half-lives of the drug (whichever is shorter) prior to the first dose of ABBV-787.
* History of documented pneumonitis that required treatment with systemic steroids within the last 6 months, nor any evidence of active pneumonitis.
* Unresolved toxicity of Grade >= 2 from prior anticancer therapy, or to levels dictated in the eligibility criteria, with the exception of alopecia.
* Known active severe or poorly controlled acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE) | Up to Approximately 3 Years
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Tolerated Dose (MTD) Based on Dose-Limiting Toxicities (DLT) | Up to approximately 28 Days
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve (AUC) of ABBV-787 | Up to Approximately 1 Year
  AUC of ABBV-787.
Maximum Observed Concentration (Cmax) of ABBV-787 | Up to Approximately 1 Year
  Cmax of ABBV-787.
Time to Cmax (Tmax) of ABBV-787 | Up to Approximately 1 Year
  Tmax of ABBV-787.
Half-life (t1/2) of ABBV-787 | Up to Approximately 1 Year
  t1/2 of ABBV-787.
Total Antibody Concentration | Up to Approximately 1 Year
  Total antibody concentration
Plasma Concentrations of Unconjugated Bromodomain and Extra-terminal Domain (BET) Degrader Payload | Up to Approximately 1 Year
  Plasma concentrations of unconjugated BET degrader payload.
Antidrug Antibody (ADA) | Up to Approximately 1 Year
  Incidence and concentration of anti-drug antibodies.
Neutralizing Antibody (nAb) | Up to Approximately 1 Year
  Incidence and concentration of neutralizing antibodies.
Percentage of Participants Achieving Complete Remission (CR) | Up to Approximately 1 Year
  CR is assessed by the European Leukemia Net (ELN). ELN defines refractory disease as the inability to attain complete remission (CR) or CR with incomplete hematologic recovery (CRi) after two courses of intensive induction treatment.
Rate of Participants Achieving CR with partial hematologic recovery (CRh) | Up to Approximately 1 Year
  Percentage of participants achieving CRh per ELN 2022.
Rate of Participants Achieving CR with incomplete hematologic recovery (CRi) | Up to Approximately 1 Year
  Percentage of participants achieving CRi per ELN 2022.
Rate of Participants Achieving Composite CR (CR, CRh, or CRi) | Up to Approximately 1 Year
  Composite CR is defined as the percentage of participants with composite CR per ELN 2022.
Rate of Participants Achieving Partial Remission (PR) | Up to Approximately 1 Year
  PR is defined as the percentage of participants with PR per ELN 2022.
Duration of Response (DOR) | Up to Approximately 1 Year
  DOR is defined for participants with CR, CRh, CRi, or PR as the time from the participant's initial response of CR, CRh, CRi, or PR per investigator review according to ELN 2022 criteria to disease progression or death of any cause, whichever occurs earlier.
Number of Participants proceeding to hematopoietic stem cell transplant (HSCT) | Up to Approximately 3 Years
  Number of participants proceeding to HSCT
Event-free Survival (EFS) | Up to Approximately 3 Years
  EFS is defined as the time from the date of the first study treatment to the date of treatment failure, or hematologic relapse from either CR, CRh, or CRi, or death from any cause, whichever occurs earlier.
Relapse free survival (RFS) | Up to Approximately 3 Years
  RFS is defined for participants achieving CR, CRh, or CRi as time from the date of achievement of remission (CR, CRh, or CRi) until the date of hematologic relapse or death from any cause.
Overall survival (OS) | Up to Approximately 3 Years
  OS is defined as time from first study treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (24):
- United States (14):
  - City of Hope /ID# 253727, Duarte, California
  - University of California Davis Health /ID# 252723, Sacramento, California
  - Yale University School of Medicine /ID# 252724, New Haven, Connecticut
  - Northwestern Memorial Hospital /ID# 252800, Chicago, Illinois
  - University of Chicago Medical /ID# 252764, Chicago, Illinois
  - University of Maryland, Baltimore /ID# 253726, Baltimore, Maryland
  - Cancer & Hematology Centers /ID# 252803, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 252515, New York, New York
  - Weill Cornell Medical College /ID# 252516, New York, New York
  - University of Pennsylvania /ID# 252789, Philadelphia, Pennsylvania
  - St. David's South Austin Medical Center /ID# 252790, Austin, Texas
  - MD Anderson Cancer Center /ID# 252514, Houston, Texas
  - Fred Hutchinson Cancer Research Center /ID# 253730, Seattle, Washington
  - Wisconsin Medical Center /ID# 252513, Milwaukee, Wisconsin
- Australia (2):
  - Monash Health - Monash Medical Centre /ID# 253841, Clayton, Victoria
  - Peter MacCallum Cancer Ctr /ID# 252517, Melbourne, Victoria
- Israel (3):
  - The Chaim Sheba Medical Center /ID# 252913, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 252914, Tel Aviv, Tel Aviv
  - Hadassah Medical Center-Hebrew University /ID# 252915, Jerusalem
- Japan (2):
  - National Cancer Center Hospital East /ID# 252519, Kashiwa-shi, Chiba
  - Yamagata University Hospital /ID# 254105, Yamagata, Yamagata
- South Korea (3):
  - Seoul National University Hospital /ID# 252916, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 253955, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 253956, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-477